CLINICAL TRIAL: NCT06161688
Title: Placebo-Controlled, Randomized Trial of Ensitrelvir (S-217622) for Viral Persistence and Inflammation in People Experiencing Long COVID (PREVAIL-LC)
Brief Title: Ensitrelvir for Viral Persistence and Inflammation in People Experiencing Long COVID
Acronym: PREVAIL-LC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Timothy Henrich (Other)
Collaborators: Shionogi Inc. (Industry)
Responsible Party: Sponsor-Investigator, Timothy Henrich, Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-38752
Record Dates: First submitted 2023-12-06; First posted 2023-12-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Long COVID; Post Acute Sequelae of COVID-19; Post-Acute COVID-19
Keywords: Antiviral; Viral Persistence
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — ensitrelvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ensitrelvir (S-217622) (Experimental): Ensitrelvir fumaric acid (S-217622) given orally 375 mg on day 1 followed by 125 mg daily for 4 additional days
  Interventions: Drug: Ensitrelvir
- Placebo (Placebo Comparator): Placebo administered orally for 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ensitrelvir — Those randomized to the experimental arm will receive Ensitrelvir, a protease inhibitor, taken orally for 5 days
  Other Names: ensitrelvir fumaric acid
  Arms: Ensitrelvir (S-217622)
Other: Placebo — Matching placebo for Ensitrelvir
  Arms: Placebo

SUMMARY:
Persistent viral infection with viral reservoirs and detection of circulating spike protein after the initial acute illness is one potential pathogenic mechanism for Long COVID. This mechanism may be susceptible to antiviral therapy that blocks viral replication, which has the potential to alleviate long COVID symptoms. This trial will study the safety and efficacy of Ensitrelvir (S-217622), an antiviral, to treat individuals with Long COVID in an adult population.

DETAILED DESCRIPTION:
The study will enroll approximately 40 participants who meet the World Health Organization (WHO) Long COVID criteria. Participants will be enrolled at a single center and randomized 1:1 to receive ensitrelvir fumaric acid (Ensitrelvir: S-217622), given orally for 5 days, or placebo. Subjects randomized to receive Ensitrelvir will take 375 mg on day 1, followed by 125 mg daily for 4 additional days. Evaluations will take place at baseline and at timepoints up to 60 days post-initiation of study drug.

ELIGIBILITY:
Inclusion Criteria (note, additional eligibility criteria not listed here will be assessed at Screening):

* ≥18 and <70 years of age at Screening.
* History of confirmed SARS-CoV-2 infection.
* Long COVID attributed to a SARS-CoV-2 infection
* At least two moderate symptoms or one severe symptom that are new or worsened since the time of a SARS-CoV-2 infection, not known to be attributable to another cause upon assessment by the PI. Symptoms must have been present for at least 60 days prior to screening and must be reported to be at least somewhat bothersome.
* Body mass index (BMI) 18 to 50 kilograms/meter squared (kg/m2), inclusive, at the time of screening.
* Participants who are of childbearing potential (CBP) and male participants with sexual partner(s) who are females of CBP must agree to use adequate contraception from study consent through 14 days after the last dose of study intervention.

Exclusion Criteria (note, additional eligibility criteria not listed here will be assessed at Screening):

* Previously received SARS-CoV-2 antiviral within 90 days prior to planned Day 0 or plan to receive such treatment before exiting the study
* Previously received COVID-19 convalescent plasma treatment within 60 days prior to planned Day 0 or plan to receive such treatment before exiting the study.
* Plans to receive any investigational or approved vaccine or booster for SARS-CoV-2 within 60 days prior to Day 0 or before Day 30 following Day 0.
* Active cardiovascular disease or recent (within 3 months) stroke.
* Recent (within 6 months) or planned major surgery.
* Currently hospitalized or recent (within 1 month) unplanned hospitalization.
* Active Hepatitis B or C infection.
* Known HIV infection.
* Severe coagulopathy (international normalized ratio ((INR) >2.0, history of hemophilia).
* Severe anemia (hemoglobin <9 grams/deciliter (g/dL)).
* Moderate or severe immunocompromise, according to the current NIH COVID-19 Treatment Guidelines as of March 6, 2023.
* History of anaphylaxis or hypersensitivity to any components of the intervention, prescription or non-prescription drugs, or food products in the past.
* Known prior diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS), preceding and not related to SARS-CoV-2 infection and not worsened since SARS-CoV-2 infection
* Pregnant, breastfeeding, or unwilling to practice birth control abide by the contraception requirements outlined in the inclusion criteria.
* Participation in a clinical trial with receipt of an investigational product within 28 days prior to Day 0.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Physical Health Summary Score from Baseline. | Baseline and Day 10
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on the PROMIS-29 scale between baseline and day 10. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). The primary outcome evaluated will be change in the Physical Health Summary Score.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Physical Health Summary Score from Baseline. | Baseline and Day 30
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on the PROMIS-29 scale between baseline and 30 days following administration. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). We will evaluate the change in the Physical Health Summary Score at these timepoints.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Mental Health Summary Score from Baseline. | Baseline and Day 10
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on the PROMIS-29 scale between baseline 10 days following administration. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). We will evaluate the change in the Mental Health Summary Score at these timepoints.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Mental Health Summary Score from Baseline. | Baseline and Day 30
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on the PROMIS-29 scale between baseline and day 30 following administration. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). We will evaluate the change in the Mental Health Summary Score at this timepoint.
Change in Quality of Life (Global Health Score) on a 100-point Visual-Analogue Scale from Baseline | Baseline and Day 10
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on self-reported score on a 100-point visual-analogue scale, where 0 represents the worst health a person can imagine and 100 represents the best health a person can imagine.
Change in Quality of Life Score (5-Item EuroQol EQ-5D-5L) Index Value Score from Baseline. | Baseline and Day 10
  5-Item EuroQol EQ-5D-5L questions assess pain/difficulty in day-to-day activities over the past week.
Change in Duke Activity Status Index (DASI) from Baseline | Baseline and Day 10
  The Duke Activity Status Index is a patient-reported estimate of functional capacity, maximal oxygen consumption (VO2 max) and maximum metabolic equivalent of tasks (METs). The DASI questionnaire produces a score between 0 and 58.2 points, which is linearly correlated with a patient's VO2 max and METs, as measured from cardiopulmonary exercise testing (CPET). It inquires about a person's ability to perform self-care, walk, climb stairs, run, do house and yard work, engage in sexual intercourse, and perform moderate recreational activities.
Change in Orthostatic Intolerance Score from Baseline | Baseline and Day 10
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on the OHQ scale between baseline and 10 days following administration. The scale assesses symptoms and their impact.
Change in World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2.0) questionnaire from Baseline | Baseline and Day 10
  The World Health Organization Disability Assessment Schedule 2.0 questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
Patient Global Impression of Change (PGIC) at D10 | Day 10
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. We will use a modified PGIC scale which has been used to study pain syndromes and has been employed in other Long COVID clinical trials. It is a common data element developed by the National Institutes of Mental Health.
Change in Everyday Cognition Form instrument from Baseline | Baseline and Day 10
  The ECog is an instrument that measures the decline in everyday cognitive and functional abilities that map to six cognitive domains, adapted specifically to describe change in abilities since having COVID. This version of the ECog questionnaire uses 41 questions to assess these domains.
Change in 6 Minute Walking Test (6MWT) from Baseline | Baseline and Day 10
  This measure will evaluate whether there is a difference between treatment with Ensitrelvir versus placebo on 6MWT performance between baseline and at 10 days following administration. The 6MWT requires an individual to walk at their normal pace for 6 minutes on a marked track (for example, a hallway). Vital signs are assessed, and the total distance covered is the primary outcome of interest.
Change in Active Stand Test from Baseline | Baseline and Day 10
  Measurements of heart rate and blood pressure measured after resting lying down, and at standardized increments for up to 10 minutes (as tolerated).
Change in Neurocognition Index (NCI) score from the CNS-VS from Baseline | Baseline and Day 10
  A neurocognitive assessment to assess motor, emotional, sensory, and cognitive function. It is available in English and Spanish and is administered using an iPad or computer.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henrich, MD, Principal Investigator — University of California, San Francisco; Michael Peluso, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF/Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No